CLINICAL TRIAL: NCT01049139
Title: Evaluation of an Intervention to Reduce Preventive Misconception in HIV Vaccine Clinical Trials
Brief Title: Preventative Misconception Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ATN 076
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-03

CONDITIONS: HIV; HIV Infections
Keywords: vaccination; HIV prevention; YMSM; youth; HIV Preventative Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No Supplemental Information (No Intervention): Participants will be administered a standard HIV vaccine trial consent form but no additional information.
- Supplemental information with 1-sided message (Experimental): Participants will be administered a standard HIV vaccine trial consent form and supplemental information with 1-sided messages (emphasizes information content related to vaccine trial randomization and unproven efficacy of vaccine).
  Interventions: Behavioral: 1-sided messages
- Supplemental information with 2-sided messages (Experimental): Participants will be administered a standard HIV vaccine trial consent form and supplemental information with 2-sided messages (acknowledges the beliefs that are at odds with the information content and seeks to neutralize those beliefs through counter-argument).
  Interventions: Behavioral: 2-sided messages

INTERVENTIONS:
Behavioral: 1-sided messages — Supplemental information with 1-sided messages (emphasizes information content related to vaccine trial randomization and unproven efficacy of vaccine).
  Arms: Supplemental information with 1-sided message
Behavioral: 2-sided messages — Supplemental information with 2-sided messages (acknowledges the beliefs that are at odds with the information content and seeks to neutralize those beliefs through counter-argument).
  Arms: Supplemental information with 2-sided messages

SUMMARY:
This study will carry out a preliminary "proof of concept" to evaluate two types of supplemental information that would serve as an adjunct to the traditional informed consent in a Human Immunodeficiency Virus (HIV) vaccine clinical trial. These will be compared to the condition where the traditional informed consent form is used alone.

Using four intervention sites, participants will be administered a standard HIV vaccine trial consent form. They will then be randomized into three conditions: 1) No supplemental information; 2) Supplemental information with 1-sided messages (emphasizes information content related to vaccine trial randomization and unproven efficacy of vaccine); and 3) Supplemental information with 2-sided messages (acknowledges the beliefs that are at odds with the information content and seeks to neutralize those beliefs through counter-argument). An interviewer-administered questionnaire (IAQ) Part 1 will be administered before the traditional HIV vaccine trial informed consent is reviewed with the participant. An IAQ Part 2 will be administered directly after the HIV vaccine trial informed consent in the control condition or after reading through the supplemental material. Debriefing interviews will be conducted with selected participants to review their understanding of the study procedures and their reactions to the supplemental materials and/or questionnaires.

The proposed research is a "proof of concept" study and is therefore not designed to test hypotheses. Consequently, formal hypothesis and related power calculations to detect certain effect sizes are not required. Instead, the goal will be to enroll an appropriate number of subjects for purpose of determining the feasibility of developing a larger study of supplemental information to be used as an adjunct to the informed consent statement in HIV vaccine clinical trials and providing related descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Not known to be HIV positive by self report; NOTE: HIV test is not a criterion for entry. Participants will be referred for HIV testing, if interested;
* A history of at least one unprotected sexual encounter involving either vaginal or anal penetration (receptive or insertive) with a male partner during the 6 months prior to enrollment;
* Between the ages of 16-19 (inclusive) at the time of informed consent/assent;
* Ability to understand both written and spoken English;
* Willing to consider enrollment into an HIV vaccine trial; and
* Gives informed consent/assent for study participation.

Exclusion Criteria:

- Anything that would impair the participant's ability to meet the study requirements (i.e. readily apparent psychiatric symptoms (hallucinations, thought disorder), visibly distraught (suicidal, homicidal, exhibiting violent behavior), intoxicated or under the influence of alcohol or other substances at the time of study enrollment*;

*NOTE: Participants cannot be visibly under the influence at the time of consent/enrollment, or during interviews.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Knowledge about phase 3 HIV vaccine clinical trials, specifically, understanding of random assignment and the unproven efficacy of the vaccine. | 7 months

SECONDARY OUTCOMES:
To carry out preliminary evaluations of potential moderators of the intervention: health literacy, numeracy, impulsivity, STI history, risk behaviors, socio-demographics (e.g., age), and health beliefs. | 7 months
Debriefing interviews with a subset of 36 participants in order to obtain feedback regarding research methodology, procedure, wording and content of the messages. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Zimet, Ph.D., Study Chair — Adolescent Trials Network
Locations (4):
- United States (4):
  - University of California at San Francisco, San Francisco, California
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland Medical School, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York

REFERENCES:
- See also: ATN Website — http://www.atnonline.org